CLINICAL TRIAL: NCT07221929
Title: Exercise-priming of CBT for Depression: the CBT+ Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-1128; R33MH129407 (NIH); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 12/19/25 (Other: UW Madison)
Record Dates: First submitted 2025-10-23; First posted 2025-10-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: cognitive behavioral therapy; CBT
MeSH Terms: conditions — Depressive Disorder, Major | interventions — RE1-silencing transcription factor; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CalmCBT (Experimental): In this arm, participants would complete 30 minutes of rest while watching a nature documentary before cognitive behavioral therapy
  Interventions: Behavioral: Rest
- ActiveCBT (Experimental): In this arm, participants would complete 30 minutes of aerobic activity before cognitive behavioral therapy, while watching the same nature documentary the CalmCBT group watches.
  Interventions: Behavioral: Aerobic Activity

INTERVENTIONS:
Behavioral: Rest — 30 minutes of rest while watching a nature documentary before cognitive behavioral therapy
  Arms: CalmCBT
Behavioral: Aerobic Activity — 30 minutes of aerobic activity before cognitive behavioral therapy, while watching the same nature documentary the CalmCBT group watches.
  Arms: ActiveCBT

SUMMARY:
This study investigates the effects of intentionally sequencing aerobic exercise immediately prior to cognitive behavioral therapy (CBT) to determine its effects on mechanisms of CBT (i.e., working alliance, behavioral activation). To assess the utility of this treatment augmentation, investigators will conduct a randomized controlled trial involving 100 adults with Major Depressive Disorder who will watch a nature documentary while either resting quietly ( 'CalmCBT') or exercising at a moderate intensity ('ActiveCBT') immediately prior to 8 weekly sessions of CBT.

DETAILED DESCRIPTION:
The overall goals of this project are to examine the efficacy of exercise priming (i.e., intentional sequencing of aerobic exercise immediately prior to cognitive behavioral therapy ['ActiveCBT']) to treat depression.

Specific aims are to 1) demonstrate the effects of exercise priming on mechanisms associated with therapy success (i.e., working alliance, behavioral activation) and 2) determine the efficacy of exercise priming for treatment of depression and strength of relationship with engagement of target CBT mechanisms.

The primary outcomes of this trial are participant-rated working alliance and change in behavioral activation each averaged across all eight sessions. Secondary outcomes include post-intervention depressive scores (Hamilton Depression Rating Scale).

For safety, suicide severity will be evaluated using the Columbia-Suicide Severity Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5) MDD, confirmed via Structured Clinical Interview for DSM-5 (SCID)
* current depressive symptoms of at least mild severity defined by a Hamilton Rating Scale of Depression (using the GRID-HAMD) score greater than or equal to 8
* EITHER not currently take any mental health medications or use other mental health treatment (e.g., behavioral, psychological) OR be on a stable mental health medication and/or treatment regimen for the past 8 weeks, and encouraged to maintain that regimen for the duration of the 8 week intervention period
* willing and safe to perform exercise based on responses on the Physical Activity Readiness Questionnaire (rules out contraindications to exercise)
* reported being CBT-naïve (as defined by never undergoing structured CBT).

Exclusion Criteria:

* reporting being currently pregnant, nursing, or planning to become pregnant during the study
* being diagnosed with current Substance Use Disorder, via the SCID
* being diagnosed with lifetime or current Psychosis, Mania, or Bipolar Disorder, via the SCID
* having class III+ obesity (BMI greater than or equal to 40)
* active suicidal ideation with specific plan and intent ('5' score on Suicidal Ideation from Columbia Suicide Severity Rating Scale [C-SSRS])
* exhibiting behavioral disturbance (e.g., aggression, mild-moderate cognitive impairment) or relationships with the study team members (e.g., therapists) that would significantly interfere with study participation, as assessed by research personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Working Alliance Inventory (WAI) - Bond subscale | data collected at each CBT session (weeks 1-8)
  The WAI-Bond subscale scores 4 items, with scores ranging from 4-28. Higher scores are stronger perceived patient-therapist bond: how the participant experiences feelings of bond (i.e., feelings of mutual trust, acceptance, and connection) with their therapist.. The Bond subscale is a primary outcome measure for this study and the total score will be analyzed as a secondary outcome.
Behavioral Activation for Depression Scale (BADS) | data collected at baseline, each CBT session (weeks 1-8), post intervention visit (week 9), week 20, week 52
  BADS is a 25-item survey, each item scored from 0 (not at all) to 6 (completely), with some items reverse scored. There are 4 sub-scales: Activation, Avoidance / Rumination, Work / School Impairment, Social Impairment. The total possible range of scores is from 0 to 150 where higher scores indicate higher behavioral activation (increased avoidance and impairment).
GRID Hamilton Rating Scale for Depression (GRID-HAMD) | baseline, post intervention visit (week 9), week 20, week 52
  The GRID-HAM-D is a 17-item clinician-completed questionnaire that will be used to rate depressive symptom severity. The questionnaire is designed for adults and is used to rate the intensity and frequency of depressive symptoms by probing mood, feelings of guilt, suicidal ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. As recommended by the Depression Rating Scale Standardization Team, Clinical Interviewers will follow the Structured Interview Guide and use GRID scoring, in which dimensions of intensity and frequency of a symptom are rated independently for each item. Higher scores reflect greater symptom severity, categorized as Normal (0-7), Mild Depression (8-13), Moderate Depression (14-18), Severe Depression (19-22), and Very Severe Depression (greater than 23).
Patient Health Questionnaire-9 (PHQ-9) | data collected at baseline, each CBT session (weeks 1-8), post intervention visit (week 9), week 20, week 52
  The PHQ-9 is a 9-item questionnaire that asks the participant to consider the last 2 weeks and score each question from 0-3 for a total possible range of scores from 0-27 where higher scores indicate increase depression.

SECONDARY OUTCOMES:
Structured Clinical Interviews for DSM-5 Disorders (SCID) | baseline, post intervention visit (week 9), week 20, week 52
  The SCID is a semi-structured interview for making diagnoses according to the diagnostic criteria published in the American Psychiatric Association's Diagnostic and Statistical Manual for Mental Disorders. Scoring on the SCID modules results in binary outcomes per each diagnostic module: either meeting criteria for a disorder or not meeting criteria for a disorder. As a secondary outcome measure, only the Major Depressive Disorder (MDD) modules of the SCID will be used. Rates of meeting MDD diagnostic criteria at baseline and post-therapy will be the primary time points used to compare remission rates between groups.
Columbia Severity Suicide Rating (CSSRS) | data collected at baseline, each CBT session (weeks 1-8), post intervention visit (week 9), week 20, week 52
  The C-SSRS will be used to assess and monitor suicide ideation and behavior. The severity of the ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with plan. Suicide behaviors are rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and non-suicidal, self-injurious behavior.
Dimensional Anhedonia Rating Scale (DARS) | Weeks 1-8 CBT sessions (repeated 3 times [before exercise/calm condition, immediately after exercise/calm condition, and after therapy]), final visit (week 9), 20-week follow up, 1-year follow up
  The DARS is a self-report measure that assesses state anhedonia across multiple domains. DARS is a 17-item survey on state anhedonia divided into four domains: hobbies, food/drink, social activities, and sensory experiences. Participants must list two activities within each of these categories that they consider their favorite and then respond to questions regarding their interest in/enjoyment of those activities on a 5-point Likert scale from "Not at all" to "Very much." During pre/post-administration, participants will be asked to respond to how they are feeling "right now."
Visual Analogue Scale (VAS) | Weeks 1-8 CBT sessions (repeated 3 times [before exercise/calm condition, immediately after exercise/calm condition, and after therapy]), final visit (week 9), 20-week follow up, 1-year follow up
  An anhedonia Visual Analog Scale [VAS] with 0 indicating 'No pleasure at all' and 100 indicating 'Greatest pleasure imaginable' will be used to measure anhedonia. In past research by the PI, correlations between the DARS and VAS were 0.49-0.69 indicating a moderate-to-strong agreement between the measures. The VAS will be used to provide a supplementary assessment of anhedonia.
Serum Brain Derived Neurotrophic Factor (BDNF) | Weeks 1, 4, and 8 CBT sessions (before exercise/calm condition, immediately after exercise/calm condition, and after therapy)
  Serum BDNF will be quantified from a standard blood draw. Blood samples collected during Visits 1, 4, and 8 will be allowed to clot for 30 minutes and then centrifuged for ten minutes at 5500 RPM and 4 ◦C. Following centrifugation, blood serum will be extracted with samples stored at -80 ◦C until BDNF analysis. Enzyme-linked immunosorbent assay (ELISA) kits will measure the concentration of total BDNF in the serum according to the manufacturer's instructions. Each blood sample will be run in duplicate and averaged.
Objective physical activity data (activPAL accelerometer) reported in minutes | Baseline, weeks 3 & 8 CBT sessions (monitors worn 1 week following each time point)
  Participants will place an activPAL on the midline of the thigh on either leg and wear the monitor during all waking hours, removing it only for water-based activities (e.g., swimming). For data to be valid, the monitor must have been worn for 20 hours on at least 4 days, including a minimum of 3 weekdays and 1 weekend day. Sleep time will be parsed out from each day's sitting/lying time automatically using PALanalysis. From these data, average minutes of sitting per day will be used to assess total sedentary time, minutes of stepping time with a cadence greater than or equal to 75 and less than 100 will be used to assess minutes of light-intensity physical activity and minutes of stepping time with a cadence greater than or equal to 100 will be used to assess minutes of moderate to vigorous physical activity (MVPA).
  Sedentary time, physical activity time and sleep time will all be recorded in minutes per day.
Objective physical activity data (activPAL accelerometer) reported in number of steps per day | Baseline, weeks 3 & 8 CBT sessions (monitors worn 1 week following each time point)
  Participants will place an activPAL on the midline of the thigh on either leg and wear the monitor during all waking hours, removing it only for water-based activities (e.g., swimming). For data to be valid, the monitor must have been worn for 20 hours on at least 4 days, including a minimum of 3 weekdays and 1 weekend day.
  Steps are recorded as cumulative number of steps per day as measured by the activPAL device.
Self-reported physical activity measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF) reported in minutes | baseline, week 4, post intervention visit (week 9), week 20, week 52
  The IPAQ is a physical activity questionnaire that inquires about average amounts of walking, moderate physical activity, vigorous physical activity, and sitting time per week. Walking and physical activity are reported in minutes per day of activity, sitting time is reported in hours per day.
36-item Short Form health survey (SF-36) | baseline, week 4, post intervention visit (week 9), week 20, week 52
  The SF-36 assesses health-related quality of life. It consists of eight scaled scores (including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher the score the less disability (i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability).
Generalized Anxiety Disorder 7 questionnaire (GAD-7) | baseline, week 4, post intervention visit (week 9), week 20, week 52
  Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for measuring generalized anxiety disorder. GAD-7 has seven items, which measure the severity of various signs of GAD according to reported response categories of: Not at all (0 points), Several days (1 point), More than half the days (2 points), and Nearly every day (3 points), with scores of 5, 10, and 15 as cut-off points for mild, moderate and severe anxiety, respectively.
Automatic Thoughts Questionnaire | baseline, weeks 1-8, post intervention visit (week 9), week 20, week 52
  The ATQ is a 30-item instrument that measures the frequency of automatic negative statements about the self. Each item is rated on the frequency of an occurrence from "not at all" to "all the time". Total scores are the sum of all 30 items, with higher totals indicating a higher level of automatic negative self-statements.
Session Evaluation Questionnaire (SEQ) | Weeks 1-8 CBT sessions
  Session Evaluation Questionnaire (SEQ) will be used to evaluate session effectiveness. This includes responses to twenty-one items in a 7-point bipolar adjective format questionnaire to assess how the client feels about each CBT session. The questionnaire assesses session depth, smoothness, positivity, and arousal. An overall score of the average of the values across each subscale will be used in this study.
Average Lyssn-generated score | Weeks 1-8 CBT sessions
  Lyssn is an AI-powered assessment platform for recording and managing session files, and all clinical interviews and therapy sessions will be recorded on the Lyssn platform. Lyssn will process the audio files from therapy sessions to generate session-level data.
  Lyssn generates metrics related to therapy effectiveness and fidelity, with individual metric scores (e.g., empathy, collaboration) ranging from 0 to 5 with higher scores indicated greater levels of the metric.
The Lam Employment Absence and Productivity Scale (LEAPS) | baseline, post intervention visit (week 9), week 20, week 52
  The LEAPS is a 10-item self-report scale that provides a measure of productivity in the workplace. Scores range from 0 to 28, with higher scores indicating higher impairment in work productivity.
The Patient Global Impression of Change scale (PGIC) | Weeks 9, 20, and 52
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. Participants respond to the prompt "Since the start of the study, my overall status is: [1] 'Very Much Improved', [2] 'Much Improved', [3] 'Minimally Improved', [4] 'No Change', [5] 'Minimally Worse', [6] 'Much Worse', or [7] 'Very Much Worse'.
REST-Q | baseline, post intervention visit (week 9), week 20, week 52
  The REST-Q is a 9-item questionnaire assessing the extent to which the participants' last night of sleep was restful or restorative. Scores range from 0-36, with higher scores indicating more restful sleep.
Emotion Regulation Questionnaire (ERQ) | baseline, post intervention visit (week 9), week 20, week 52
  The ERQ is a 10-item scale measuring emotional regulation on a 7-point scale for each question (total range: 7-70). Higher scores indicate increased use of emotion regulation strategies.
Rumination Reflection Questionnaire (RRQ) | baseline, post intervention visit (week 9), week 20, week 52
  The RRQ is a 24-item questionnaire assessing levels of rumination. Each item is scored 1-5 (total scores ranging 24-120). Higher scores indicate higher levels of rumination.
Working Alliance Inventory (WAI) - Total | data collected at each CBT session (weeks 1-8)
  The WAI scores 12 items from 1-7 in 3 domains: Tasks (4-28), Goals (4-28), Bond (4-28). Total possible range of scores from 12-84. In all domains higher scores are stronger perceived working alliance. The Bond subscale is a primary outcome measure. The total score and the two other subscales, Tasks and Goals, will be analyzed as secondary outcomes.

OTHER OUTCOMES:
Health history questions | Baseline, any changes reported at week 9 for medication and service use
  Health history and service use will be self-reported. In addition, participants will be asked to list their current medications.
Demographic questionnaire | Baseline
  Demographic characteristics including age, sex, race, education, marital status, occupational status, and household income will be recorded or measured to characterize the sample.
Adverse Childhood Experience Survey (ACES) | Baseline
  The ACES consists of 16 questions pertaining to the respondents' first 18 years of life. Participants respond with yes or no regarding if a childhood adverse event occurred. Adverse events questions are grouped by categories. Participants are scored for each event category they are exposed to with scores ranging from 0 (unexposed) to 7 (exposed to all categories).
World Health Organization Disability Assessment Schedule (WHODAS) | Baseline, post intervention visit (week 9)
  A 12-item subscale of the WHODAS is used at baseline to record any difficulties due to health conditions. Each item is scored 0-4, with higher scores indicate higher level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Meyer, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Questionnaire data will be shared with the NIMH Data Archives (NDA).
Supporting Information: ICF
Time Frame: IPD will be available one year after the final NIMH NDA data upload.
Access Criteria: Individuals who submit request to access for IPD to NIMH NDA may be able to access the data.
URL: https://nda.nih.gov/nda/access-data-info

REFERENCES:
- [Background] Meyer JD, Kelly SJE, Gidley JM, Lansing JE, Smith SL, Churchill SL, Thomas EBK, Goldberg SB, Abercrombie HC, Murray TA, Wade NG. Protocol for a randomized controlled trial: exercise-priming of CBT for depression (the CBT+ trial). Trials. 2024 Oct 7;25(1):663. doi: 10.1186/s13063-024-08495-x. PMID 39375728